CLINICAL TRIAL: NCT04783740
Title: Validity and Reliability of Turkish Version of The Working Memory Questionnaire
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, MSc, Research Assistant, Kutahya Health Sciences University
Other Study IDs: KutahyaHSU
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-03

CONDITIONS: Working Memory; The Working Memory Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to determine the Turkish validity and reliability of ''The Working Memory Questionnaire'' developed by Dr. Vallat-Azouvi.

DETAILED DESCRIPTION:
Working Memory refers to the temporary storage and exchange of information required for complex tasks such as language, understanding, learning, and reasoning. Working memory deficits are worse in people with advanced age and low education. In addition, working memory is impaired in children with traumatic brain injury, stroke, Alzheimer's disease, and attention deficit hyperactivity disorder. The aim of this study is to determine the Turkish version, validity, and reliability of ''The Working Memory Questionnaire''. 300 health people will include in the study. In order to determine the reliability of the scale, the intraclass correlation coefficient (ICC) will be used to determine the level of the relationship between the results of the first and second measurements. Cronbach's alpha coefficient will be used for the homogeneity of the questions in the scale. For construct validity, the correlation coefficient will be used to determine the agreement between the Turkish Version of Cognitive Failures Questionnaire and The Working Memory Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being an individual between the ages of 18-50

Exclusion Criteria:

* Having a neurological and mental illness

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Individuals living in Turkey
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The Working Memory Questionnaire | 15 minute
  The Working Memory Questionnaire has been designed by Dr. Vallat-Azouvi at el. specifically to assess everyday life difficulties related to working memory failures. It consists of 30 statements rated on a 5-point Likert-type scale ranging from "not at all" to "extremely". WMQ is consists of 3 subscales, there are storage, attention, and executive domains.The total score ranges from 0-120 points. Higher scores correspond to more self-identified difficulties

SECONDARY OUTCOMES:
Turkish Version Cognitive Failures Questionnaire | 12 minute
  The Cognitive Failures Questionnaire (CFQ) is a self-report questionnaire to assess failures of perception, motor function, and memory. CFQ is consists of 25 items and 5 points Likert-type scale. The total score is ranges from 0-100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Caner AKSOY, PhD, Study Director — Kutahya Health Sciences University; İsmail SARAÇOĞLU, PhD, Principal Investigator — Kutahya Health Sciences University; Lütfiye AKKURT, MSc, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No